CLINICAL TRIAL: NCT04325191
Title: Melatonin and Salt on Blood Vessel Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1534734
Record Dates: First submitted 2020-03-19; First posted 2020-03-27 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Cardiovascular Risk Factor
Keywords: Vascular Health; Melatonin; Dietary Sodium; Blood Pressure
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: This is a randomized crossover design trial.
Who Masked: Participant
Masking Description: Participant will not know if they are receiving the melatonin or placebo pills.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Salt and Melatonin (Experimental): Subjects will consume sodium pills throughout the day achieving a total of 6900 mg sodium/day (4600 mg of sodium from pills and 2300 mg from diet) and will supplement with 10 mg (single dose) of melatonin at night.
  Interventions: Dietary Supplement: Melatonin
- High Salt and Placebo (Placebo Comparator): Subjects will consume sodium pills throughout the day achieving a total of 6900 mg sodium/day (4600 mg of sodium from pills and 2300 mg from diet) and will supplement with a lactose placebo (single dose) at night.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Daily consumption of a high sodium diet and melatonin for 10 days
  Arms: High Salt and Melatonin
Other: Placebo — aily consumption of a high sodium diet and placebo for 10 days
  Arms: High Salt and Placebo

SUMMARY:
Increased dietary sodium causes increases in oxidative stress and damages blood vessels. Americans eat more than the recommended amount of sodium. Melatonin is a powerful endogenous antioxidant that has reduced oxidative stress levels in clinical and healthy populations. This study will investigate whether melatonin can attenuate the negative effects of sodium on blood vessels.

DETAILED DESCRIPTION:
Americans consume on average double the recommended amount of sodium established by organizations such as the American Heart Association and the Dietary Guidelines for Americans. Excess dietary sodium damages the inside of our blood vessels in a process known as endothelial dysfunction. This reduces the ability of blood vessels to dilate as much. This type of dysfunction can lead to the development of cardiovascular disease. Animal and human studies have identified one potential mechanism linking high sodium consumption and endothelial dysfunction; that is oxidative stress. Furthermore, high dietary sodium consumption has been shown to increase blood pressure reactivity in animal studies. Melatonin is a powerful endogenous antioxidant that has reduced oxidative stress levels in clinical and healthy populations. Melatonin has been shown to attenuate sympathetic responses, but research is limited. Whether supplementation of melatonin can offset the deleterious effects of a high sodium diet is unknown. Thus, the purpose of this study is to investigate the effect of melatonin supplementation compared to a placebo on markers of oxidative stress and blood vessel function in healthy young adults that consume a 10-day high sodium diet. Our hypotheses are that: 1) melatonin will reduce oxidative stress levels and restore blood vessel function and 2) melatonin will reduce the sympathetic nerve response to high sodium consumption.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* normal blood pressure

Exclusion Criteria:

* hypertension
* heart disease
* diabetes
* kidney disease
* renal impairment
* cancer
* obese (BMI ≥30)
* sleep disorder
* use of tobacco products
* pregnant or breastfeeding
* take any medications for the above conditions
* endurance trained athletes
* night shift worker
* melatonin or antioxidant consumption for the previous 3 months
* use of selective serotonin reuptake inhibitors

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Conduit artery endothelial-dependent function | Day 10
  Assessed by brachial artery flow mediated dilation (FMD)
Microvascular function | Day 10
  Assessed by Near Infrared Spectroscopy (NIRS)

SECONDARY OUTCOMES:
Blood pressure reactivity | Day 10
  Assessed by the change in blood pressure during Handgrip Exercise and Cold Pressor test from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Shannon L Lennon, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States